CLINICAL TRIAL: NCT03794921
Title: Leveraging Technology to Address Access and Adherence to Conventional Hospital-Based Pulmonary Rehabilitation in Veterans With COPD
Brief Title: COPD Access to Pulmonary Rehabilitation Intervention
Acronym: CAPRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F2855-R; I01RX002855 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2019-01-07 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: COPD
Keywords: Pulmonary Rehabilitation; Technology-Mediated; Web-Based Intervention; Physical Activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: As the primary aim, the investigators propose a RCT to study the efficacy of a web-based, pedometer-mediated physical activity intervention to increase physical activity in persons with COPD who would benefit from but cannot access conventional pulmonary rehabilitation, compared to usual care. The investigators anticipate that 120 subjects will be randomized 1:1 to either the intervention or usual care.
Who Masked: Outcomes Assessor
Masking Description: Study staff communicating randomization assignments to subjects will be different from study staff conducting follow-up outcome assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Patients referred to conventional PR or eligible for PR but declined or cannot access. Using a standardized script at the randomization phone call, study staff will deliver verbal instructions to slowly and steadily increase one's walking and exercise each week. Participants will be asked to perform exercise of moderate intensity for at least 30 minutes on most days of the week, defined as a dyspnea level of 4-5 on the Borg scale and taking 1-2 minutes to recover. Use of the Borg rating scale for dyspnea will be reviewed with each participant. Exercise is defined as planned PA, outside of activities performed as part of one's daily routine. Exercise can be walking in the community or using exercise equipment at a local gym. Adapted written materials reinforce the verbal instructions. Participants will receive this 45-page spiral-bound book with information about aerobic and strength training exercises.
- Every Step Counts Intervention (Experimental): Patients referred to conventional PR or eligible for PR but declined or cannot access. After randomization to ESC, participants will be mailed detailed instructions about the website. They will be asked to wear the lightweight, unobtrusive pedometer every day, except while asleep or showering/bathing, during the 12-week intervention period. Subjects will be instructed to upload their date and time-stamped step-count data to the study website at least weekly. Each week, the study computer will run the goal calculation algorithm and provide each participant with his/her daily step-count goal for the week. The week's step-count goal will be displayed on each subject's personal study web page. Participants will be instructed to exercise and reach their individualized step-count goals with walking of moderate intensity for at least 30 minutes on most days of the week, defined as a dyspnea level of 4-5 on the Borg scale and taking 1-2 minutes to recover.
  Interventions: Other: Every Step Counts

INTERVENTIONS:
Other: Every Step Counts — Pedometer coupled to a website that provides step-count goals, feedback, education, motivation, and social support.
  Arms: Every Step Counts Intervention

SUMMARY:
Persons with COPD have significant functional disability but cannot access rehabilitative treatment at hospital-based conventional pulmonary rehabilitation (PR) programs. This project will determine whether an Internet-mediated, pedometer-based walking program can increase physical activity in persons with COPD who qualify for but cannot access PR, compared to usual care. This proposal has high potential to deliver an immediate solution to a pressing clinical need. The proposed research addresses Rehabilitation R&D Service's current priority area of improving disabled Veterans' health-related quality of life by reducing disease burden and maximizing functional recovery.

DETAILED DESCRIPTION:
Conventional pulmonary rehabilitation (PR) programs are highly effective and the standard of care in patients with chronic obstructive pulmonary disease (COPD). PR faces two significant problems: (1) most patients with COPD who would benefit from PR cannot access it, and 2) there is no effective long-term strategy to maintain physical activity (PA) and benefits after completing PR. The investigators propose a randomized controlled trial (RCT) to test the efficacy of a technology-mediated intervention to increase PA in persons with COPD who qualify for but cannot access conventional, hospital-based PR. COPD is a leading cause of death in the United States; an estimated 16 million Americans have COPD. Despite maximal medical therapy, patients with COPD characteristically experience breathlessness, which leads to a downward spiral of sedentary behavior, physical inactivity, deconditioning, and functional disability. Low physical activity is associated with poor outcomes in COPD--increased risk of acute exacerbations, hospitalizations, and death, independent of lung function. The Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines recommend regular PA for all patients with COPD. Conventional, supervised PR programs clearly reduce breathlessness, and improve health-related quality of life (HRQL) and exercise capacity. However, PR programs face significant challenges of access and adherence. The investigators developed Every Step Counts (ESC), a technology-mediated intervention based on the Behavioral Theory of Self-Regulation, to target sedentary behavior, promote PA, and alleviate deconditioning. ESC couples a website with a pedometer to directly monitor step counts. The website provides individualized step-count goals, iterative feedback, education on disease self-management, motivation, and an online community of social support. In two randomized studies in Veterans with COPD, the investigators demonstrated ESC's safety, feasibility, and efficacy to increase PA. Accessible via the internet and available at any time from home, ESC could be an ideal low-cost platform to address the limitations of conventional PR. The investigators hypothesize that ESC may be an efficacious strategy to promote PA in the many patients who cannot attend a PR program.

Primary Aim 1: Determine the efficacy of a web-based intervention, ESC, to increase PA (measured directly with an accelerometer and a questionnaire that assesses intensity), compared to usual care, in persons with COPD who are referred to or eligible for conventional PR but who cannot access it.

Secondary Aim 2: Estimate the effect of the ESC intervention on (a) exercise self-efficacy, (b) HRQL, (c) dyspnea, (d) depression, and (e) risk of acute exacerbations and COPD-related hospitalizations, compared to usual care.

All study visits are performed either in-person or remotely starting September, 2021.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, greater than or equal to 40 years of age
* Clinical diagnosis of COPD defined as either a ratio of FEV1 to forced vital capacity (FVC) < 0.70 or chest CT evidence of emphysema or prior documentation of FEV1/FVC ratio of < 0.7 and clinical evidence of COPD

  * defined as 10 pack-year cigarette smoking history
  * dyspnea
  * or on bronchodilators
* Have declined participation in or cannot access a conventional pulmonary rehabilitation program
* Medical clearance from healthcare provider to participate in an exercise program
* Have access to a computer with Internet connection, a USB port or Bluetooth capability, and Windows XP/Vista/7/8/10 or higher, or Mac OSX 10.5 or higher operating system, or willing to come to VA Medical Center to use study computers
* Competent to provide informed consent
* Willingness to make return visits and be available by telephone for duration of study

Exclusion Criteria:

* COPD exacerbation in the previous 1 month
* Inability to ambulate with or without assistance (if remote)
* On supplemental oxygen (if remote)
* Use of walking assistive device (if remote)
* Inability to complete questionnaires
* Inability to collect at least 7 of 10 days of baseline step counts
* Participation in a pulmonary rehabilitation program at time of screening or within the previous 3 months
* Participation in another exercise-related research study at time of screening
* Plans to participate in an exercise-related research study in the next 3 months
* Average baseline step counts of greater than or equal to 10,000 steps per week

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Physical Activity measured as Daily Step Count | 12 weeks
  Daily Step Count directly measured with a monitoring device.

SECONDARY OUTCOMES:
Exercise Self-Regulatory Efficacy | 12 weeks
  Assessed by the Exercise Self-Regulatory Efficacy Scale questionnaire. 16-item questionnaire. Participants indicate their confidence level from 0% (not at all confident) to 100% (highly confident).
Health-Related Quality of Life using a disease specific questionnaire | 12 weeks
  Assessed by the St. George's Respiratory Questionnaire. The investigators will use the Total Score and the 3 Domains of Activity, Symptoms, and Impacts. Scores range from 0 to 100, with lower scores representing better health related quality of life.
Shortness of Breath rating as perceived by the participant | 12 weeks
  Shortness of Breath is one outcome measured in 2 ways. It will be assessed by the University of California, San Diego (UCSD) Shortness of Breath (SOB) Questionnaire and the modified Medical Research Council scale. The UCSD SOB Questionnaire contains 24 items with scores ranging from 0 to 120. The modified Medical Research Council (mMRC) dyspnea scale ranges from 0 to 4, with higher numbers representing more shortness of breath.
Healthcare Utilization represented by number of Acute Exacerbations and Hospitalizations over timeframe | 12 weeks
  Acute Exacerbation and Hospitalization History. Assessment of total number of acute exacerbations (AEs) and hospitalizations over the timeframe of 12 weeks and 6 months is based on both self-report and medical chart review.
Amount of Depression experienced by the participant | 12 weeks and 6 months
  Depression measured by the Beck's Depression Inventory-II questionnaire. 21-items. Scores range with 0 to 63 with higher scores representing greater severity of depression.

OTHER OUTCOMES:
Health Utilities | 12 weeks
  EuroQoL 5-Dimension Health Questionnaire (EQ-5D) Health Utilities. 2 pages assesses 5 dimensions with visual analog scale. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. The EQ VAS (EQ visual analogue scale) records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labeled 'Best imaginable health state' and 'Worst imaginable health state'.
Number of participants who enroll in Conventional Pulm Rehab after participating in the research study | 12 weeks
  Numbers will be assessed by self-report and chart review.
COPD Knowledge | 12 weeks
  Bristol COPD Knowledge Questionnaire. 13-items that usually takes between 10 and 20 minutes to complete. Percent of questions scored correctly is assessed and range from 0 to 100 %.
Sleepiness | 12 weeks
  Epworth Sleepiness Scale. 8 questions, each on a scale of 0-3. Minimum score is 0 and maximum score is 24.
  0-5 Lower Normal Daytime Sleepiness 6-10 Higher Normal Daytime Sleepiness 11-12 Mild Excessive Daytime Sleepiness 13-15 Moderate Excessive Daytime Sleepiness 16-24 Severe Excessive Daytime Sleepiness
Social Support | 12 weeks
  MOS Social Support Survey. 18 items with scores ranging from 0 to 100, with higher scores representing greater social support.
Brief Pain Inventory | 12 weeks
  Pain Severity Score (8 items) is calculated by adding the scores for questions 2, 3, 4 and 5 and then dividing by 4. This gives a severity score out of 10. Pain Interference Score is calculated by adding the scores for questions 8a, b, c, d, e, f and g and then dividing by 7. This gives an interference score out of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn L. Moy, MD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Datasets meeting VA standards for disclosure to the public will be made available within 1 year of publication.
  * A local privacy officer will certify that a dataset contains no Protected Health Information (PHI), Personally Identifiable Information (PII), or VA Sensitive Information prior to release outside VA.
  * Final data sets will be maintained locally on a secure server or comparable data storage appliance inside the VA network until enterprise-level resources become available for long-term storage and access.
  The PI will create de-identified, study-specific datasets. Investigators requesting a copy of a dataset will sign a Letter of Agreement or a Data Use Agreement. A local privacy officer will certify that a dataset contains no PHI, PII, or VA Sensitive Information prior to release outside VA.